CLINICAL TRIAL: NCT00003128
Title: A Phase III Trial of Ifosfamide (NSC #109274) Versus Ifosfamide Plus Paclitaxel (NSC #125973) in Patients With Advanced, Persistent or Recurrent Carcinosarcoma (Mixed Mesodermal Tumors) of the Uterus
Brief Title: Ifosfamide With or Without Paclitaxel in Treating Patients With Advanced, Refractory, or Recurrent Cancer of the Uterus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065891; GOG-0161; ECOG-G0161
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2004-05

CONDITIONS: Sarcoma
Keywords: stage III uterine sarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma; uterine carcinosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Filgrastim; Ifosfamide; Paclitaxel

INTERVENTIONS:
Biological: filgrastim
Drug: ifosfamide
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether ifosfamide alone is more effective than ifosfamide plus paclitaxel in treating patients with cancer of the uterus.

PURPOSE: Randomized phase III trial to compare the effectiveness of ifosfamide with or without paclitaxel in treating patients with advanced, refractory, or recurrent cancer of the uterus.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the addition of paclitaxel to ifosfamide improves length of survival, progression free interval and response rate when compared to ifosfamide alone in patients with advanced, refractory or recurrent carcinosarcoma (mixed mesodermal tumors) of the uterus.
* Determine the toxicity of ifosfamide with paclitaxel in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to GOG performance status (GOG 0-1 vs GOG 2-3) and randomized to one of two treatment arms.

* Arm I: Patients receive ifosfamide IV daily for 3 days every 21 days.
* Arm II: Patients receive paclitaxel IV on day 1 and ifosfamide IV on days 1-3 every 21 days. Filgrastim (G-CSF) is given subcutaneously beginning on day 4 until granulocyte count is greater than 2,000/mm3. Paclitaxel therapy may precede or be given concurrently with ifosfamide.

Treatment for both arms continues for a maximum of 8 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, then every 6 months for an additional 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 166 patients (83 per arm) will be accrued for this study within approximately 5.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III or IV, refractory, or recurrent heterologous or homologous carcinosarcoma (mixed mesodermal tumors) of the uterus
* Must not be amenable to curative-intent therapy
* Must have measurable disease consisting of abdominal, pelvic, chest or other masses that can be defined in at least 2 dimensions by palpation, x-ray, MRI, computed tomography or ultrasound

  * If measured by MRI, computed tomography or ultrasound, the lesion must have a minimal tumor measurement of 1 cm

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Albumin at least 3 g/dL
* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No history of congestive heart failure
* No unstable angina
* No myocardial infarction within the past 6 months

Other:

* No septicemia
* No severe infection
* No acute hepatitis
* No gastrointestinal bleeding
* At least 5 years since any other invasive malignancy except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for carcinosarcoma of the uterus

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 6 weeks since radiotherapy for current malignancy
* At least 3 months since radiotherapy if delivered to site of measurable disease

Surgery:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 1997-11; Primary Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard D. Homesley, MD, Study Chair — Gynecologic Oncology Network; Higinia R. Cardenes, MD, PhD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (17):
- United States (17):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Tufts - New England Medical Center, Boston, Massachusetts
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth Medical School, Lebanon, New Hampshire
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Abramson Cancer Center at University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - Scott and White Hospital, Temple, Texas

REFERENCES:
- [Result] Homesley HD, Filiaci V, Markman M, Bitterman P, Eaton L, Kilgore LC, Monk BJ, Ueland FR; Gynecologic Oncology Group. Phase III trial of ifosfamide with or without paclitaxel in advanced uterine carcinosarcoma: a Gynecologic Oncology Group Study. J Clin Oncol. 2007 Feb 10;25(5):526-31. doi: 10.1200/JCO.2006.06.4907. PMID 17290061